CLINICAL TRIAL: NCT04023058
Title: Stress Echo for Ischemic Mitral Valve Surgery
Acronym: SURVIVE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy director for science, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2/2019
Record Dates: First submitted 2019-06-30; First posted 2019-07-17 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Mitral Regurgitation
Keywords: ischemic mitral regurgitation; mitral surgery; stress echo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CABG/increasing MR (No Intervention): non-massive IMR with increasing IMR during exercise - CABG only
- CABG+mitral surgery (MS)/increasing MR (Experimental): non-massive IMR with increasing IMR during exercise - CABG+ mitral surgery
  Interventions: Procedure: Mitral surgery
- CABG/non-increasing MR (No Intervention): non-massive IMR non-increasing IMR during exercise - CABG only
- CABG+MS/non-increasing MR (Experimental): non-massive IMR non-increasing IMR - CABG+ mitral surgery
  Interventions: Procedure: Mitral surgery
- Control 1 (Other): massive IMR at rest without increasing during exercise - CABG+ mitral surgery
  Interventions: Procedure: Mitral surgery
- Control 2 (Other): massive IMR at rest with increasing during exercise - CABG+ mitral surgery
  Interventions: Procedure: Mitral surgery

INTERVENTIONS:
Procedure: Mitral surgery — Guidelines approved mitral surgery
  Arms: CABG+MS/non-increasing MR; CABG+mitral surgery (MS)/increasing MR; Control 1; Control 2

SUMMARY:
Comparison patients with CABG alone vs. CABG+mitral surgery with non-massive ischaemic mitral regurgitation (IMR) depending on stress echo data.

DETAILED DESCRIPTION:
Chronic ischaemic mitral regurgitation (IMR) is a frequent complication of coronary artery disease (CAD), and is associated with a poor prognosis and outcome. The role of concomitant mitral valve surgery for IMR in patients undergoing coronary artery bypass grafting (CABG) remains controversial. After myocardial infarction IMR is associated with poor outcome and prognosis with double mortality rates, it reduces survival following surgical or percutaneous revascularization. However, there is no consensus on the cut-off value of IMR. The thresholds to define severe secondary mitral regurgitation are need to be evaluated with regards to their impact on prognosis after mitral valve intervention. The European guidelines is defined effective regurgitant orifice (ERO)-0.2 cm2 and regurgitant volume (RV)-30ml, as the threshold for severe IMR, because of severe prognosis of this group. Whereas American guidelines are defined it as ERO-0.4 cm2 and RV-60ml, as it was no evidence to impact intervention on the IMR with ERO-0.2 cm2 and RV-30ml. Partly it's explained by the dynamic nature of the secondary MR. About 30% of patients from the group with non-massive regurgitation at rest, have dramatically increasing it during exercise. However, some patient have not changes or decreasing IMR during exercise and, probably, they have not such a negative impact on the hemodynamic by IMR. The pervious comparative studies, that were the base for recommendations did not differ the patients with and without changes IMR during exercise. The current guidelines doesn't support the stress echo (SE) exams before operation for assessing necessity in mitral valve operation. It's due to lack of information that prove of influence for survival after surgery depending on IMR dynamic parameters.

IMR study hypothesis: Stress echocardiography data, including ERO, RV, pulmonary pressure (PA) pressure, beta-lines - B-lines, contractile reserve, could be indications for mitral valve intervention in patient with CAD and chronic secondary mitral regurgitation, undergoing CABG. The patients of the group with non-massive (ERO-0.2 cm2 and RV-30ml) IMR have positive effect by mitral surgery if they have increasing IMR during exercise test. The group with massive IMR (ERO≥0.4 cm2 and RV≥60 ml) will be better according clinic, echo, stress echo results in comparison with non-massive non-operated subgroup.

Aim: To assess the value of stress echo testing for ischemic mitral surgery indication in patients undergoing CABG.

Inclusion criteria for all projects are:

1. Age > 18 years
2. IMR, ERO≥0.2 cm2 and RV≥30 ml.
3. Indication for CABG

Exclusion criteria for all projects are:

1. Unwillingness to give informed consent and to enter a regular follow-up program.
2. Contraindications for stress echo.

Methods and design:

1. In a prospective multicenter international randomized study, we will recruit patients whom CABG is planned.
2. Conventional transthoracic echo. Patients will include into two groups:

   Group 1 - "Non-massive IMR" - ERO-0.2-0.39 cm2, and RV-30-59ml. Group 2 - "Massive IMR" - ERO≥0.4 cm2 and RV≥60 ml.
3. Randomization of Group 1 (surgery/non-surgery).
4. Exercise stress echocardiography of all the patients (Group 1 and Group 2). regional wall motion abnormality (RWMA), ejection fraction (EF), end diastolic volume (EDV), end systolic volume (ESV), contractile reserve, B-lines, ERO, RV, PA pressure at rest and during stress.
5. 1-year clinical outcomes
6. 1-year transthoracic echo data.
7. 1-year stress echocardiography data.
8. 3-year clinical outcomes
9. 3-year transthoracic echo data.
10. 3-year stress echocardiography data. Primary end-points: death, myocardial infarction, new hospital readmission, heart transplant, ventricular assist device implantation, aborted sudden death, pulmonary oedema (MACE).

Secondary end-points: physical capacity (changes in Watts, minutes of stress echocardiography), EDV, left atrium volume, EF at rest and during SE, ERO, RV, PA pressure, B-lines, contractile reserve at rest and during exercise in comparison with pre-operative data.

Expected results. Group 1, CABG - subgroup, CABG+mitral surgery subgroup. It's expected the improvement of physical capacity (changes in Watts, minutes of stress echocardiography), EDV, left atrium volume, EF at rest and during SE, ERO, RV, PA pressure, B-lines, contractile reserve at rest and during exercise in comparison with pre-operative data in CABG+mitral surgery subgroup already in 1-year follow-up. It's expected the improvement of physical capacity (changes in Watts, minutes of stress echo), EDV, left atrium volume, EF at rest and during stress echo, ERO, RV, PA pressure, B-lines, contractile reserve at rest and during exercise in comparison with CABG-subgroup already in 1-year follow-up. It's expected that more pronounce changes will be in CABG+mitral surgery subgroup with previously increasing IMR. The worst results are expected in CABG-subgroup with previously increasing IMR during exercise. There will be clarified which parameters would be more correlate with the clinic improvement (contractile reserve, B-lines, ERO etc). We expected reduced MACE till 3 year in CABG+mitral surgery subgroup with increasing IMR in comparison with CABG-subgroup with increasing IMR.

Group 2, The group with massive IMR (ERO≥0.4 cm2 and RV≥60 ml) will be better according clinic, echo, stress echo results in comparison with CABG-subgroup with increasing IMR from group 1. There will be clarified which parameters would be more correlate with the clinic improvement (contractile reserve, B-lines, ERO etc).

ELIGIBILITY:
Inclusion Criteria:

* Ischemic MR, ERO≥0.2 cm2 and RV≥30 ml.
* Indication for CABG

Exclusion Criteria:

* Unwillingness to give informed consent and to enter a regular follow-up program.
* Contraindications for SE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
myocardial infarction | during 3 year
  myocardial infarction
all-cause death | during 3 year
  all-cause death
new hospital readmission | during 3 year from including
  new hospitalization
re-operation | during 3 year
  percutaneous coronary intervention, coronary bypass surgery, heart transplant
cardiac death | during 3 year
  cardiac death

SECONDARY OUTCOMES:
physical capacity | Change from Baseline of physical capacity in Watts at 12 months, at 3 years
  Change in Watts during stress test
end diastolic volume of left ventricle | Change from Baseline of end diastolic volume of left ventricle at 12 months, at 3 years
  Change in milliliters by echocardiography
left atrium volume | Change from Baseline of left atrium volume at 12 months, at 3 years
  Change in milliliters by echocardiography
ejection fraction at rest and during stress echo | Change from Baseline of ejection fraction at 12 months, at 3 years
  Change in percent by echocardiography at rest and at the peak of exercise during stress test
effective regurgitant orifice | Change from Baseline at 12 months, at 3 years
  Change in centimeter square of mitral effective regurgitant orifice by echocardiography
right ventricle size | Change from Baseline at 12 months, at 3 years
  Change in centimeter of right ventricle by echocardiography
pulmonary artery pressure pressure | Change from Baseline at 12 months, at 3 years
  Change in mm Hg of pulmonary pressure by echocardiography
B-lines | Change from Baseline at 12 months, at 3 years
  counts of B-lines during by stress echocardiography
Contractile reserve | Change from Baseline at 12 months, at 3 years
  Change in contractile reserve by stress echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shmatov, MD, PhD, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- St. Petersburg State University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 year

DOCUMENTS (1):
  • Informed Consent Form (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04023058/ICF_000.pdf